CLINICAL TRIAL: NCT02469246
Title: A Phase 3b, Randomized, Double-Blind, Switch Study to Evaluate F/TAF in HIV-1 Infected Subjects Who Are Virologically Suppressed on Regimens Containing ABC/3TC
Brief Title: Switch Study to Evaluate F/TAF in HIV-1 Infected Adults Who Are Virologically Suppressed on Regimens Containing ABC/3TC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-311-1717; 2015-000871-28 (EudraCT Number)
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: HIV-1 Infection
Keywords: HIV; HIV-1 Positive; Virologically-Suppressed
MeSH Terms: interventions — emtricitabine tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- F/TAF (Double-Blind) (Experimental): F/TAF + ABC/3TC placebo + allowed 3rd antiretroviral (ARV) agent for 96 weeks
  After Week 96, participants will continue to take their blinded study drug and attend visits every 12 weeks until treatment assignments have been unblinded.
  Interventions: Drug: F/TAF; Drug: ABC/3TC Placebo; Drug: 3rd ARV agent
- ABC/3TC (Double-Blind) (Active Comparator): ABC/3TC + F/TAF placebo + allowed 3rd ARV agent for 96 weeks
  After Week 96, participants will continue to take their blinded study drug and attend visits every 12 weeks until treatment assignments have been unblinded.
  Interventions: Drug: ABC/3TC; Drug: F/TAF Placebo; Drug: 3rd ARV agent
- Open-Label F/TAF (Experimental): After the unblinding visit, in countries where F/TAF FDC is not commercially available, participants (except in certain countries such as the UK) will be given the option to receive open-label F/TAF (200/10 mg or 200/25 mg) FDC and attend study visits every 12 weeks until it becomes commercially available, or until Gilead terminates the study in that country.
  Interventions: Drug: F/TAF

INTERVENTIONS:
Drug: F/TAF — 200/10 mg FDC tablet (with boosted 3rd ARV agents) or 200/25 mg FDC tablet (with unboosted 3rd ARV agents) administered orally once daily
  Other Names: Descovy®
  Arms: F/TAF (Double-Blind); Open-Label F/TAF
Drug: ABC/3TC — 600/300 mg FDC tablets administered orally once daily
  Arms: ABC/3TC (Double-Blind)
Drug: ABC/3TC Placebo — Tablets administered orally once daily
  Arms: F/TAF (Double-Blind)
Drug: F/TAF Placebo — Tablets administered orally once daily
  Arms: ABC/3TC (Double-Blind)
Drug: 3rd ARV agent — An allowed 3rd ARV agent of the participant's pre-existing regimen may include one of the following boosted ARV agents: ritonavir boosted lopinavir (LPV/r), atazanavir (ATV) + ritonavir (RTV), ATV + cobicistat (COBI) or ATV/COBI FDC, darunavir (DRV) + RTV, DRV+COBI or DRV/COBI FDC; or, one of the following unboosted ARV agents: efavirenz (EFV), rilpivirine (RPV), raltegravir (RAL), dolutegravir (DTG), maraviroc (MVC), or nevirapine (NVP).
  Arms: ABC/3TC (Double-Blind); F/TAF (Double-Blind)

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of switching abacavir/lamivudine (ABC/3TC) fixed-dose combination (FDC) tablets to emtricitabine/tenofovir alafenamide (F/TAF) FDC tablets versus maintaining ABC/3TC in human immunodeficiency virus type 1 (HIV-1) infected adults who are virologically suppressed on regimens containing ABC/3TC.

ELIGIBILITY:
Key Inclusion Criteria:

* The ability to understand and sign a written informed consent form
* On antiretroviral regimen containing ABC/3TC FDC in combination with one 3rd agent for ≥ 6 consecutive months prior to screening
* Plasma HIV-1 RNA levels < 50 copies/mL for ≥ 6 months preceding the screening visit (measured at least twice using the same assay) and without experiencing two consecutive HIV-1 RNA above detectable levels after achieving a confirmed (two consecutive) HIV-1 RNA below detectable levels on the current regimen in the past year
* Plasma HIV-1 RNA should be < 50 copies/mL at the screening visit
* Normal ECG
* Estimated glomerular filtration rate (GFR) ≥ 50 mL/min according to the Cockcroft Gault formula for creatinine clearance
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Females of childbearing potential and males must agree to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 30 days following the last dose of study drug

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen (HBsAg) positive
* Individuals experiencing decompensated cirrhosis
* Individuals receiving ongoing treatment with bisphosphonate to treat bone disease (eg, osteoporosis)
* Pregnant or lactating females
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the investigator to potentially interfere with study compliance
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1 Visit
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval
* Medications excluded due to the potential for interaction with emtricitabine (FTC), TAF, ABC or 3TC

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (80):
- United States (34):
  - Spectrum Medical Group, Phoenix, Arizona
  - Pacific Oaks Medical Group, Beverly Hills, California
  - University of California San Diego (UCSD), La Jolla, California
  - Anthony Mills, MD, Inc., Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Highland Hospital - Alameda Health System, Oakland, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Capial Medical Associates, Washington D.C., District of Columbia
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Gary J. Richmond,M.D.,P.A., Fort Lauderdale, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Atlanta ID Group, Atlanta, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Be Well Medical Center, Berkley, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The KC CARE Clinic, Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - AIDS Arms, Inc, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Peter Shalit, MD, Seattle, Washington
- Belgium (2):
  - UZ Gent, Ghent
  - Centre Hospitalier Universitaire CHU Sart Tilman Liege, Liège
- Canada (4):
  - Clinique medicale l'Actuel, Montreal
  - Maple Leaf Research, Toronto
  - Spectrum Health, Vancouver
  - Vancouver ID Research and Care Centre Society, Vancouver
- Hvidovre Hospital, Copenhagen, Denmark
- France (5):
  - CHU - Groupe Saint-Andre, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - C.H.U. de Nantes, Nantes
  - CHR Orleans la Source, Orléans
  - Chu Tours, Tours
- Germany (8):
  - ICH Study Center Hamburg, Bielefeld
  - Medizinische Universitatsklinik, Bonn
  - Klinikum der Universitaet Koln, Cologne
  - Universitatsklinikum Essen, Essen
  - Johann Wolfgang Goethe-University Hospital, Frankfurt
  - ifi-Studien und Projekte GmbH an der Asklepiosklinik St. Georg, Hamburg
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum München, Munich
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - Saint James's Hospital, Dublin
- Italy (6):
  - University of Brescia, Brescia
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Fondazione IRCCS San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Roma
  - Ospedale Amedeo di Savoia - Specializzato Malattie infettive, Torino
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan
  - Hope Clinical Research Inc, San Juan
- Spain (6):
  - Bonaventura, Badalona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Costa Del Sol, Málaga
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (9):
  - Birmingham Heartlands Hospital, Birmingham
  - Barts Health NHS Trust, London
  - Chelsea and Westminster Hospital, London
  - Imperial College, London
  - Kings College Hospital NHS Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - Royal Free Hospital, London
  - St. George's Hospital, London
  - Manchester Centre for Sexual Health, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Winston A, Post FA, DeJesus E, Podzamczer D, Di Perri G, Estrada V, Raffi F, Ruane P, Peyrani P, Crofoot G, Mallon PWG, Castelli F, Yan M, Cox S, Das M, Cheng A, Rhee MS. Tenofovir alafenamide plus emtricitabine versus abacavir plus lamivudine for treatment of virologically suppressed HIV-1-infected adults: a randomised, double-blind, active-controlled, non-inferiority phase 3 trial. Lancet HIV. 2018 Apr;5(4):e162-e171. doi: 10.1016/S2352-3018(18)30010-9. Epub 2018 Feb 20. PMID 29475804
- [Result] Gupta SK, Post FA, Arribas JR, Eron JJ Jr, Wohl DA, Clarke AE, Sax PE, Stellbrink HJ, Esser S, Pozniak AL, Podzamczer D, Waters L, Orkin C, Rockstroh JK, Mudrikova T, Negredo E, Elion RA, Guo S, Zhong L, Carter C, Martin H, Brainard D, SenGupta D, Das M. Renal safety of tenofovir alafenamide vs. tenofovir disoproxil fumarate: a pooled analysis of 26 clinical trials. AIDS. 2019 Jul 15;33(9):1455-1465. doi: 10.1097/QAD.0000000000002223. PMID 30932951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Europe. The first participant was screened on 29 June 2015. The last study visit occurred on 13 March 2019.
Pre-assignment Details: 626 participants were screened.
Groups:
- F/TAF: Double-Blind Phase: Emtricitabine/tenofovir alafenamide (F/TAF) (200/10 mg) fixed-dose combination (FDC) tablet (with boosted 3rd antiretroviral (ARV) agent) or F/TAF (200/25 mg) FDC tablet (with unboosted 3rd ARV agent) + abacavir/lamivudine (ABC/3TC) placebo tablet once daily for 96 weeks, and continued blinded treatment until unblinding. [Allowed boosted 3rd ARV agents: ritonavir boosted lopinavir (LPV/r), atazanavir (ATV) + ritonavir (RTV), ATV + cobicistat (COBI) or ATV/COBI FDC, darunavir (DRV) + RTV, DRV+COBI or DRV/COBI FDC; Allowed unboosted 3rd ARV agents: efavirenz (EFV), rilpivirine (RPV), raltegravir (RAL), dolutegravir (DTG), maraviroc (MVC), or nevirapine (NVP)].
  Open-Label Extension: After the unblinding visit, in countries where F/TAF FDC was not commercially available, participants (except in certain countries) were given the option to receive the open-label F/TAF FDC until it became commercially available, or until Gilead terminated the study in that country.
- ABC/3TC: Double-Blind Phase: ABC/3TC (600/300 mg) FDC tablet + F/TAF placebo tablet once daily + allowed 3rd ARV agent for 96 weeks, and continued blinded treatment until unblinding. (Allowed boosted 3rd ARV agents: LPV/r, ATV + RTV, ATV + COBI or ATV/COBI FDC, DRV + RTV, DRV+COBI or DRV/COBI FDC; Allowed unboosted 3rd ARV agents: EFV, RPV, RAL, DTG, MVC, or NVP)
  Open-Label Extension: After the unblinding visit, in countries where F/TAF FDC was not commercially available, participants (except in certain countries) were given the option to receive the open-label F/TAF FDC until it became commercially available, or until Gilead terminated the study in that country.
Period: Double-Blind Phase
Arm/Group | F/TAF | ABC/3TC
Started | 285 | 282
Completed | 218 | 226
Not Completed | 67 | 56
Not completed — Randomized and Never Treated | 5 | 6
Not completed — Adverse Event | 12 | 9
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 2 | 1
Not completed — Investigator's Discretion | 8 | 8
Not completed — Non-Compliance with Study Drug | 3 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrew Consent | 25 | 25
Not completed — Lost to Follow-up | 9 | 5
Period: Open-Label Extension (OLE)
Arm/Group | F/TAF | ABC/3TC
Started | 6 (Only participants in countries where F/TAF was not commercially available were eligible for the OLE.) | 5 (Only participants in countries where F/TAF was not commercially available were eligible for the OLE.)
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who received at least one dose of study drug. Participants were grouped according to the treatment they actually received.
Groups:
- F/TAF: F/TAF (200/10 mg) FDC tablet (with boosted 3rd ARV agent) or F/TAF (200/25 mg) FDC tablet (with unboosted 3rd ARV agent) + ABC/3TC placebo tablet once daily for 96 weeks
- ABC/3TC: ABC/3TC (600/300 mg) FDC tablet + F/TAF placebo tablet once daily + allowed 3rd ARV agent for 96 weeks
- Total: Total of all reporting groups
Arm/Group | F/TAF | ABC/3TC | Total
Number analyzed (Participants) | 280 | 276 | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.4) | 51 (9.3) | 51 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 61 | 101
  Male | 240 | 215 | 455
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 35
  Not Hispanic or Latino | 264 | 257 | 521
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 5 | 10
  Black | 64 | 66 | 130
  White | 205 | 199 | 404
  Other | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 6 | 10
  Canada | 9 | 8 | 17
  Denmark | 4 | 3 | 7
  France | 18 | 17 | 35
  Germany | 20 | 19 | 39
  Ireland | 9 | 8 | 17
  Italy | 26 | 17 | 43
  Spain | 32 | 34 | 66
  Sweden | 3 | 4 | 7
  United Kingdom | 50 | 59 | 109
  United States | 105 | 101 | 206
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 278 | 273 | 551
  ≥ 50 copies/mL | 2 | 3 | 5
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 703 (298.7) | 727 (275.2) | 715 (287.3)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/µL | 0 | 1 | 1
  ≥ 50 to < 200 cells/µL | 0 | 0 | 0
  ≥ 200 to < 350 cells/µL | 20 | 16 | 36
  ≥ 350 to < 500 cells/µL | 56 | 38 | 94
  ≥ 500 cells/µL | 204 | 221 | 425
HIV Disease Status [Count of Participants; unit: Participants]
  Asymptomatic | 201 | 201 | 402
  Symptomatic HIV Infection | 31 | 24 | 55
  AIDS | 47 | 50 | 97
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug. Participants were grouped according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 88.6 | 92.4
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; The analysis purpose of the primary efficacy endpoint was to assess the noninferiority of switching to F/TAF+3rd Agent relative to maintaining treatment with ABC/3TC+3rd Agent; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% confidence interval (CI) approach, with a non-inferiority margin of 10%; p = 0.15, Fisher Exact; Difference in Percentages = -3.8, 95.002% CI 2-sided [-8.9 to 1.1] — The difference in percentages and its 95.002% CI were calculated based on an unconditional exact method using 2 inverted 1-sided tests

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 82.1 | 88.4
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; The analysis purpose of this efficacy endpoint was to assess the non-inferiority of switching to F/TAF+3rd Agent relative to maintaining treatment with ABC/3TC+3rd Agent; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% CI approach, with a non-inferiority margin of 4%; p = 0.042, Fisher Exact; Difference in Percentages = -6.3, 95% CI 2-sided [-12.3 to -0.3] — The difference in percentages and its 95% CI were calculated based on an unconditional exact method using 2 inverted 1-sided tests

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 1.8 | 0.7
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% CI approach, with a non-inferiority margin of 4%; p = 0.45, Fisher Exact; Difference in Percentages = 1.1, 95.002% CI 2-sided [-1.0 to 3.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 96 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 2.5 | 1.1
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% CI approach, with a non-inferiority margin of 4%; p = 0.34, Fisher Exact; Difference in Percentages = 1.4, 95% CI 2-sided [-1.0 to 4.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 48 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 85.7 | 87.3
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; The analysis purpose of this efficacy endpoint was to assess the noninferiority of switching to F/TAF+3rd Agent relative to maintaining treatment with ABC/3TC+3rd Agent; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% CI approach, with a non-inferiority margin of 10%; p = 0.62, Fisher Exact; Difference in Percentages = -1.6, 95% CI 2-sided [-7.4 to 4.2] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 20 Copies/mL at Week 96 as Determined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 20 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 280 | 276
percentage of participants | 80.4 | 86.2
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; [analysis description as in outcome 5, analysis 1]; Test type: Non-Inferiority — Non-inferiority was assessed using a 2-sided exact 95% CI approach, with a non-inferiority margin of 10%; p = 0.069, Fisher Exact; Difference in Percentages = -5.9, 95% CI 2-sided [-12.2 to 0.4] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 249 | 254
cells/µL | -30 (152.3) | 2 (171.2)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.026, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = -32, 95% CI 2-sided [-61 to -4] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

8. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 229 | 238
cells/μL | -29 (160.7) | 10 (178.2)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.013, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = -39, 95% CI 2-sided [-70 to -8] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

9. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Hip Dual-Energy X-Ray Absorptiometry (DXA) Analysis Set (all participants who are randomized and have received at least one dose of study drug, and have nonmissing baseline hip BMD values) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 231 | 236
percent change | 0.246 (2.2914) | 0.086 (2.3315)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.40, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = 0.179, 95% CI 2-sided [-0.240 to 0.598] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

10. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 213 | 221
percent change | 0.169 (2.7277) | 0.021 (2.7212)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.53, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = 0.165, 95% CI 2-sided [-0.348 to 0.678] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

11. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (all participants who are randomized and have received at least one dose of study drug, and have nonmissing baseline spine BMD values) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 232 | 240
percent change | 0.081 (3.0051) | -0.052 (3.7550)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.63, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = 0.151, 95% CI 2-sided [-0.465 to 0.767] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

12. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | F/TAF | ABC/3TC
Number analyzed (Participants) | 217 | 225
percent change | 0.178 (3.8881) | 0.235 (4.3066)
Statistical Analysis 1: Comparison: F/TAF vs ABC/3TC; Test type: Superiority; p = 0.89, ANOVA — P-value was adjusted by the third agent stratum (boosted protease inhibitors vs. others); Difference in LSM = -0.056, 95% CI 2-sided [-0.825 to 0.713] — Difference in LSM and its 95% CI were adjusted by the third agent stratum (boosted protease inhibitors vs. others)

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (maximum duration: 168 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- F/TAF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the F/TAF group, who received F/TAF (200/10 mg) FDC tablet (with boosted 3rd ARV agent) or F/TAF (200/25 mg) FDC tablet (with unboosted 3rd ARV agent) + ABC/3TC placebo tablet once daily.
- ABC/3TC (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the ABC/3TC group, who received ABC/3TC (600/300 mg) FDC tablet + F/TAF placebo tablet once daily + allowed 3rd ARV agent.
- Open-Label F/TAF From F/TAF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the F/TAF group and received F/TAF (200/10 mg or 200/25 mg) FDC tablet once daily.
- Open-Label F/TAF From ABC/3TC: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the ABC/3TC group and received F/TAF (200/10 mg or 200/25 mg) FDC tablet once daily.
Arm/Group | F/TAF (Double-Blind Phase) | ABC/3TC (Double-Blind Phase) | Open-Label F/TAF From F/TAF | Open-Label F/TAF From ABC/3TC
All-Cause Mortality (participants affected / at risk) | 5/280 | 0/276 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 55/280 | 32/276 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 190/280 | 199/276 | 1/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF (Double-Blind Phase) (N=280) | ABC/3TC (Double-Blind Phase) (N=276) | Open-Label F/TAF From F/TAF (N=6) | Open-Label F/TAF From ABC/3TC (N=5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Acute hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 2 | 0 | 0
Viral myocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Viral load increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Substance use (Social circumstances) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | F/TAF (Double-Blind Phase) (N=280) | ABC/3TC (Double-Blind Phase) (N=276) | Open-Label F/TAF From F/TAF (N=6) | Open-Label F/TAF From ABC/3TC (N=5)
Diarrhoea (Gastrointestinal disorders) | 30 | 37 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 11 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 10 | 0 | 0
Fatigue (General disorders) | 21 | 15 | 0 | 0
Bronchitis (Infections and infestations) | 19 | 14 | 0 | 0
Gastroenteritis (Infections and infestations) | 11 | 15 | 0 | 0
Influenza (Infections and infestations) | 12 | 15 | 0 | 0
Nasopharyngitis (Infections and infestations) | 57 | 49 | 0 | 1
Rhinitis (Infections and infestations) | 7 | 6 | 0 | 1
Syphilis (Infections and infestations) | 15 | 5 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 36 | 46 | 0 | 0
Urinary tract infection (Infections and infestations) | 13 | 18 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 29 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 31 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 14 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 15 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 31 | 25 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 30 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 14 | 17 | 0 | 0
Hypertension (Vascular disorders) | 15 | 15 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02469246/Prot_000.pdf
  • Statistical Analysis Plan: Week 48 (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT02469246/SAP_001.pdf
  • Statistical Analysis Plan: Final Analysis (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT02469246/SAP_002.pdf